CLINICAL TRIAL: NCT02948686
Title: Clinical Evaluation of Different Application Strategies When Using a Universal Adhesive System in Class V Cavities
Brief Title: Different Application Strategies When Using Ambar Universal in Class V Cavities
Acronym: AUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFFAMBAR2016
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: dentin bonding agents; tooth sensitivity; composite resin restoration
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SET (Self-Etching) (Active Comparator): 55 teeth will receive restorations using Self-Etching Application Strategy
  Interventions: Other: Self-Etching Application Strategy
- SEE (Selective Enamel Etching) (Experimental): 55 teeth will receive restorations using Enamel Etching Application Strategy
  Interventions: Other: Enamel Etching Application Strategy
- SETT (Self-Etching, more time) (Experimental): 55 teeth will receive restorations using Self Etching with Extended time Application Strategy
  Interventions: Other: Self Etching with Extended time Application Strategy
- SETL (Self-Etching, more layers) (Experimental): 55 teeth will receive restorations using Self Etching with Extended layers number Strategy
  Interventions: Other: Self Etching with Extended layers number Strategy

INTERVENTIONS:
Other: Self-Etching Application Strategy — In Group SET, the adhesive system Ambar Universal will be used in 55 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 10 seconds in the cavity, will be air-dried during 5 seconds, brushed again during 10 seconds, air-dried during 10 seconds and activated during 10 seconds with LED light; After applying the adhesive, the restorations will be made with composite resin Opallis (FGM, Joinville, Brazil), and evaluated every 6 months for pain assessment, shape, staining or recurrent caries, using scores.
  Arms: SET (Self-Etching)
Other: Enamel Etching Application Strategy — In Group SEE, 37% phosphoric acid will be applied during 15 seconds, only in enamel in 55 teeth. This acid will be removed using water, the cavity will be air-dried, and then, the adhesive system Ambar Universal will be brushed during 10 seconds in the cavity, will be air-dried during 5 seconds, brushed again during 10 seconds, air-dried during 10 seconds and activated during 10 seconds with LED light; After applying the adhesive, the restorations will be made with composite resin Opallis (FGM, Joinville, Brazil), and evaluated every 6 months for pain assessment, shape, staining or recurrent caries, using scores.
  Arms: SEE (Selective Enamel Etching)
Other: Self Etching with Extended time Application Strategy — In Group SETT, the adhesive system Ambar Universal will be used in 55 teeth, in the self-etching mode. The adhesive system will be brushed during 20 seconds in the cavity, will be air-dried during 5 seconds, brushed again during 20 seconds, air-dried during 10 seconds and activated during 10 seconds with LED light; After applying the adhesive, the restorations will be made with composite resin Opallis (FGM, Joinville, Brazil), and evaluated every 6 months for pain assessment, shape, staining or recurrent caries, using scores
  Arms: SETT (Self-Etching, more time)
Other: Self Etching with Extended layers number Strategy — In Group SETL, the adhesive system Ambar Universal will be used in 55 teeth, in the self-etching mode. The adhesive system will be brushed during 10 seconds in the cavity, will be air-dried during 5 seconds, brushed again during 10 seconds, air-dried during 5 seconds, brushed again during 10 seconds, air-dried during 5 seconds, brushed again during 10 seconds, air-dried during 5 seconds, and activated during 10 seconds with LED light; After applying the adhesive, the restorations will be made with composite resin Opallis (FGM, Joinville, Brazil), and evaluated every 6 months for pain assessment, shape, staining or recurrent caries, using scores
  Arms: SETL (Self-Etching, more layers)

SUMMARY:
Treatment clinical trial, randomized, controled, parallel, double-blinded, with four groups, that aims to evaluate the best application strategy when using a new Universal Adhesive system, Ambar Universal (FGM, Joinville, Brazil). Volunteers will be selected and recruited,following inclusion criteria and pre-established exclusion. All volunteers will be informed and sign a term of clarification and consent. 38 enrolled patients will receive four Class V dental restorations, made in four different ways, one from each experimental group, using the same universal self-etching adhesive system, which is the tested material in this study. Non-carious cervical lesions will receive the applied adhesive system in 4 different protocols separated by groups. Group Self Etching (SET) (control): no conditioning, the adhesive system will be used in 55 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 10 seconds in the cavity, will be air-dried during 5 seconds, brushed again during 10 seconds, air-dried during 10 seconds and activated during 10 seconds with Light Emission Diode (LED) light; Group SEE (Selective enamel etching): 37% phosphoric acid will be applied during 15 seconds, only in enamel in 55 teeth. This acid will be removed using water, the cavity will be air-dried, and then, the adhesive will be applied according to the manufacturer's instructions, as described in group SET; Group SETT (Self-Etching with extended time): Similar to Group SET, but during the 2 applications, the adhesive systems will be brushed during 20 seconds, and not during 10 seconds as described in Group SET; Group SETL (Self-Etching with extended number of layers): The adhesive system will be applied as describe in Group SET, but the researchers will apply 4 layers, and not 2 layers, as described in Group SET. After applying the adhesive, the restorations will be made with composite resin, and evaluated every 6 months for pain assessment, shape, staining or recurrent caries, using scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

DETAILED DESCRIPTION:
This is a Treatment clinical trial, randomized, controlled, parallel, double-blinded, with four groups, that aims to evaluate the best application strategy when using a new Universal Adhesive system, Ambar Universal (FGM, Joinville, Brazil). Volunteers will be selected and recruited,following inclusion criteria and pre-established exclusion. All volunteers will be informed and sign a term of clarification and consent. All 38 enrolled patients will receive Class V dental restorations, made in four different ways, one from each experimental group, using the same universal self-etching adhesive system, which is the tested material in this study. All patients must have at only 20 teeth in function, must have at only 4 non carious cervical lesions (NCCL), in different teeth, that need restoration. Those lesions must be non carious, must be more than 1 mm deep, should have exposed dentin, and must have at only 50% of margins in enamel. Teeth should not present periodontal mobility. Firstly, the patient will be anesthetized locally with 3% Mepivacaine solution, followed by prophylaxis with pumice powder and water. All cavities will be washed and dried after these procedures for optimal selection of color, using a color scale. Then, the rubber dam isolation of the teeth to be restored will be held. Non-carious cervical lesions will receive the applied adhesive system in 4 different protocols separated by groups. Group SET (control): no conditioning, the adhesive system will be used in 55 teeth, according to the manufacturer's instructions, in the self-etching mode. The adhesive system will be brushed during 10 seconds in the cavity, will be air-dried during 5 seconds, brushed again during 10 seconds, air-dried during 10 seconds and activated during 10 seconds with LED light; Group SEE (Selective enamel etching): 37% phosphoric acid will be applied during 15 seconds, only in enamel in 55 teeth. This acid will be removed using water, the cavity will be air-dried, and then, the adhesive will be applied according to the manufacturer's instructions, as described in group SET; Group SETT: Similar to Group SET, but during the 2 applications, the adhesive systems will be brushed during 20 seconds, and not during 10 seconds as described in Group SET; Group SETL: The adhesive system will be applied as describe in Group SET, but the researchers will apply 4 layers, and not 2 layers, as described in Group SET. After applying the adhesive, the restorations will be made with composite resin Opallis (FGM, Joinville, Brazil), and evaluated every 6 months for pain assessment, shape, staining or recurrent caries, using scores. To determine in which group each tooth will be enrolled, the authors will randomize the teeth.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have at only 20 teeth in function, must have at only 4 non carious cervical lesions (NCCL), in different teeth, that need restoration. Those lesions must be non carious, must be more than 1 mm deep, should have exposed dentin, and must have at only 50% of margins in enamel. Teeth should not present periodontal mobility.

Exclusion Criteria:

* Volunteers with periodontal disease; with gingival bleeding; use of anti-inflammatory drugs in the last 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Restoration Loss | Four years
  It will be evaluated the increase in the number of losses of dental restorations in the period of four years, verified by periodic visual clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of remaining restorations in the different groups.

SECONDARY OUTCOMES:
Marginal Pigmentation | Four years
  It will be evaluated the increase in the number of dental restorations with marginal pigmentation in the period of four years, verified by periodic clinical visual examination (6/6 months) based on the statement of difference of at least 25% in the amount of stained restorations in the different groups.
Post-Operative Hypersensitivity | Four years
  It will be evaluated the increase in the number of dental restorations with dentin hypersensitivity in the period of four years, verified by periodic clinical examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with dentin hypersensitivity in the different groups.
Secondary Caries | Four years
  It will be evaluated the increase in the number of dental restorations with secondary caries in the period of four years, verified by periodic radiographic examination (6/6 months) based on the statement of difference of at least 25% in the amount of restorations with secondary caries in the different groups.

CONTACTS AND LOCATIONS:
Overall Officials: MARCOS O BARCELEIRO, DDS, PHD, Study Director — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense - School of Dentistry, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pashley DH, Tay FR. Aggressiveness of contemporary self-etching adhesives. Part II: etching effects on unground enamel. Dent Mater. 2001 Sep;17(5):430-44. doi: 10.1016/s0109-5641(00)00104-4. PMID 11445211
- [Background] Perdigao J, Kose C, Mena-Serrano AP, De Paula EA, Tay LY, Reis A, Loguercio AD. A new universal simplified adhesive: 18-month clinical evaluation. Oper Dent. 2014 Mar-Apr;39(2):113-27. doi: 10.2341/13-045-C. Epub 2013 Jun 26. PMID 23802645
- [Background] Erhardt MC, Cavalcante LM, Pimenta LA. Influence of phosphoric acid pretreatment on self-etching bond strengths. J Esthet Restor Dent. 2004;16(1):33-40; discussion 41. doi: 10.1111/j.1708-8240.2004.tb00448.x. PMID 15259541
- [Background] Erickson RL, Barkmeier WW, Latta MA. The role of etching in bonding to enamel: a comparison of self-etching and etch-and-rinse adhesive systems. Dent Mater. 2009 Nov;25(11):1459-67. doi: 10.1016/j.dental.2009.07.002. Epub 2009 Aug 7. PMID 19665220
- [Background] Torii Y, Itou K, Nishitani Y, Ishikawa K, Suzuki K. Effect of phosphoric acid etching prior to self-etching primer application on adhesion of resin composite to enamel and dentin. Am J Dent. 2002 Oct;15(5):305-8. PMID 12537339
- [Background] Van Landuyt KL, Peumans M, De Munck J, Lambrechts P, Van Meerbeek B. Extension of a one-step self-etch adhesive into a multi-step adhesive. Dent Mater. 2006 Jun;22(6):533-44. doi: 10.1016/j.dental.2005.05.010. Epub 2005 Nov 21. PMID 16300826
- [Background] da Costa TR, Ferri LD, Loguercio AD, Reis A. Eighteen-month randomized clinical trial on the performance of two etch-and-rinse adhesives in non-carious cervical lesions. Am J Dent. 2014 Dec;27(6):312-7. PMID 25707085
- [Background] Lopes LS, Calazans FS, Hidalgo R, Buitrago LL, Gutierrez F, Reis A, Loguercio AD, Barceleiro MO. Six-month Follow-up of Cervical Composite Restorations Placed With a New Universal Adhesive System: A Randomized Clinical Trial. Oper Dent. 2016 Sep-Oct;41(5):465-480. doi: 10.2341/15-309-C. Epub 2016 Jul 5. PMID 27379834
- [Background] Swift EJ Jr, Perdigao J, Heymann HO, Wilder AD Jr, Bayne SC, May KN Jr, Sturdevant JR, Roberson TM. Eighteen-month clinical evaluation of a filled and unfilled dentin adhesive. J Dent. 2001 Jan;29(1):1-6. doi: 10.1016/s0300-5712(00)00050-6. PMID 11137632
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Int Dent J. 2007 Oct;57(5):300-2. doi: 10.1111/j.1875-595x.2007.tb00136.x. No abstract available. PMID 17992913
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Dalton Bittencourt D, Ezecelevski IG, Reis A, Van Dijken JW, Loguercio AD. An 18-months' evaluation of self-etch and etch & rinse adhesive in non-carious cervical lesions. Acta Odontol Scand. 2005 Jun;63(3):173-8. doi: 10.1080/00016350510019874. PMID 16191912